CLINICAL TRIAL: NCT06499168
Title: CD10 as a Prognostic and Predictive Factor to Neoadjuvant Chemotherapy Response in Locally Advanced Breast Cancer
Brief Title: Predicting Response to Neoadjuvant Chemotherapy in Locally Advanced Breast Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Rehab Osama Abdelmaboud, assistant lecturer, Assiut University
Other Study IDs: response to NAC in LABC
Record Dates: First submitted 2024-07-06; First posted 2024-07-12 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Locally Advanced Breast Cancer
Keywords: response, neoadjuvant chemotherapy, breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Formalin fixed paraffin embedded tissue specimen of the baseline TCNB of locally advanced breast cancer will be obtained from pathology laboratory, Pathology Department, Assiut University.
  * Histological diagnosis of H&E stained sections will be confirmed.
  * Immunohistochemical staining for CD10 .
  * Baseline clinicopathological features of patients who received neoadjuvant chemotherapy will be collected from patients' records.
  * Correlation between CD10 expression and the baseline clinicopathological features with the response to neoadjuvant chemotherapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- groups: LABC patients who will receive neoadjuvant chemotherapy before surgery.
  Interventions: Drug: neoadjuvant chemotherapy: anthracycline based chemotherapy and taxans before surgery

INTERVENTIONS:
Drug: neoadjuvant chemotherapy: anthracycline based chemotherapy and taxans before surgery — In locally advanced breast cancer patients who will receive neoadjuvant chemotherapy formalin fixed paraffin embedded tissue specimen of the baseline TCNB of locally advanced breast cancer will be obtained from pathology laboratory, Pathology Department, Assiut University.
  * Histological diagnosis of H&E stained sections will be confirmed.
  * Immunohistochemical staining for CD10 .
  * Baseline clinicopathological features of patients who will receive neoadjuvant chemotherapy will be collected from patients' records.
  * Correlation between CD10 expression and the baseline clinicopathological features with the response to neoadjuvant chemotherapy.

SUMMARY:
Female breast cancer is the second leading cause of global cancer incidence in 2022 and the fourth leading cause of cancer mortality worldwide. Breast cancer (BC) remains the most prevalent cancer diagnosis among women; nevertheless, considerable advancements in diagnostics and treatment approaches have significantly enhanced patient outcomes. In locally advanced cases, primary systemic chemotherapy is often indicated, and the choice of treatment is influenced by the evaluation of routine prognostic and predictive factors.

Neoadjuvant chemotherapy (NCT) has emerged as a valuable approach to enhance the quality of life ,disease-free and overall survival for early and locally advanced BC patients Approximately 30% of BC cases achieve a pathological complete response (pCR) following NCT. Unfortunately, proper quantification of estrogen- and progesterone receptors (ER and PR), human epidermal growth factor receptor-2 (HER2/Neu) and proliferation markers are insufficient to predict chemosensitivity of some breast tumors , so the identification of these cases during routine pathological examination of biopsy specimens could be especially useful in planning the oncotherapeutic strategy for proper patient management.

CD10, has recently gained attention as an independent diagnostic and prognostic marker in various solid tumors with significant metastatic potential. This molecule has been shown to play a role in cell adhesion, migration, and extracellular matrix remodelling.

A strong CD10 expression has been linked to hormone receptor negativity and HER-2/neu overexpression in breast cancer. Moreover, the dynamics of stromal CD10 expression undergo changes during neoadjuvant anthracycline-based chemotherapy.

Recent research, has presented compelling data indicating that CD10 expression may serve as a predictive marker for the impact of neoadjuvant chemotherapy in breast cancer patients.

DETAILED DESCRIPTION:
Formalin fixed paraffin embedded tissue specimen of the baseline TCNB of locally advanced breast cancer will be obtained from pathology laboratory, Pathology Department, Assiut University.

* Histological diagnosis of H&E stained sections will be confirmed.
* Immunohistochemical staining for CD10 .
* Baseline clinicopathological features of patients who will receive neoadjuvant chemotherapy will be collected from patients' records.
* Correlation between CD10 expression and the baseline clinicopathological features with the response to neoadjuvant chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients above 18 years
* Pathologically proven breast carcinoma
* Locally advanced breast cancer

Exclusion Criteria:

* Patients below 18 years.
* Patients with metastatic disease
* Patients with second primary cancer
* Patients ineligible for chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Data Record of the patients will be reviewed for the following:
  Clinical features:
  * Age
  * Menopausal status
  * Family history
  * contraception
  * Comorbidities.
  Pathological features:
  * Histological type of breast carcinoma
  * Grade
  * Lymphovascular invasion(LVI)
  * Ductal carcinoma insitu
  * TNM stage.
  * ER, PR, HER2 and Ki67.
  Immunohistochemistry (IHC):
  CD 10 expression by IHC staining
  Type of Neoadjuvant CTH received:
  * AC (Adriamycin -cyclophosphamide)
  * taxans
  Number of cycles
  Response to neoadjuvant Chemotherapy:
  Follow up :
  Follow up of the patient during the course of treatment including evaluation of the patients by examination cycle by cycle till surgery to assess the adverse events and to evaluate the clinical response in addition to preoperative MRI or breast sonomamography.
  Follow up after finishing the course of treatment by imaging and examination every 3 months for 2 years.
Sampling Method: Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
The response to neoadjuvant chemotherapy in locally advanced breast cancer in relation to CD10 expression | 6 months

SECONDARY OUTCOMES:
progression free survival (PFS) | 2 years
  the average length of time after the start of treatment in which a person is alive and their cancer does not grow or spread
Overall survival (OS) | 2 years
  the average length of time patients are alive after diagnosis or the start of treatment